CLINICAL TRIAL: NCT05651321
Title: A Series of Studies on the Impact of Taste-aware Intelligent Analysis of Oral Nutritional Supplements on Patients' Nutritional Strategies
Brief Title: Studies on the Impact of Taste-aware Intelligent Analysis of Oral Nutritional Supplements
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: ONSTaste2.0
Record Dates: First submitted 2022-12-05; First posted 2022-12-15 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2022-12

CONDITIONS: Cancer- and Cancer Treatment-Related Conditions; Stroke
MeSH Terms: conditions — Neoplasms; Stroke

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- stroke patients: Participants were tested for different taste perception thresholds using a three-point difference test, with samples materials for basic taste stimuli were used, i.e. reference substances tartaric/citric acid (acidic), quinine hydrochloride/caffeine (bitter), anhydrous sodium chloride (salty), sucrose (sweet), and quercetin/alum (astringent) were used to prepare different tastes and concentrations of liquids. The subjects will then evaluate the appearance (color, texture), taste, flavor, and texture of the six different flavored enteral nutrition preparations. The subjects will then perform manual sensory evaluation of the appearance (color, texture), odor, taste, texture, and other properties of the 6 different flavored enteral nutrition preparations.
  Interventions: Other: Samples materials of basic taste stimuli and enteral nutrition preparations
- cancer patients: Participants were tested for different taste perception thresholds using a three-point difference test, with samples materials for basic taste stimuli were used, i.e. reference substances tartaric/citric acid (acidic), quinine hydrochloride/caffeine (bitter), anhydrous sodium chloride (salty), sucrose (sweet), and quercetin/alum (astringent) were used to prepare different tastes and concentrations of liquids. The subjects will then evaluate the appearance (color, texture), taste, flavor, and texture of the six different flavored enteral nutrition preparations. The subjects will then perform manual sensory evaluation of the appearance (color, texture), odor, taste, texture, and other properties of the 6 different flavored enteral nutrition preparations.
  Interventions: Other: Samples materials of basic taste stimuli and enteral nutrition preparations
- healthy people: Participants were tested for different taste perception thresholds using a three-point difference test, with samples materials for basic taste stimuli were used, i.e. reference substances tartaric/citric acid (acidic), quinine hydrochloride/caffeine (bitter), anhydrous sodium chloride (salty), sucrose (sweet), and quercetin/alum (astringent) were used to prepare different tastes and concentrations of liquids. The subjects will then evaluate the appearance (color, texture), taste, flavor, and texture of the six different flavored enteral nutrition preparations. The subjects will then perform manual sensory evaluation of the appearance (color, texture), odor, taste, texture, and other properties of the 6 different flavored enteral nutrition preparations.
  Interventions: Other: Samples materials of basic taste stimuli and enteral nutrition preparations

INTERVENTIONS:
Other: Samples materials of basic taste stimuli and enteral nutrition preparations — Samples materials of basic taste stimuli were used, i.e. reference substances tartaric/citric acid (acidic), quinine hydrochloride/caffeine (bitter), anhydrous sodium chloride (salty), sucrose (sweet), and quercetin/alum (astringent) and six different flavored enteral nutrition preparations.

SUMMARY:
The goal of this observational study is to test the taste perception threshold and palatability interval of different populations and the difference in taste perception between tumor and stroke patients and healthy people by combining manual sensory evaluation and electronic bionic sensory and investigate the taste perception characteristics and demand of enteral nutrition preparations such as Fortimel in tumor and stroke patients, and the difference in taste perception of enteral nutrition preparations with healthy people by combining manual sensory evaluation and electronic bionic sensory. Participants were tested for different taste perception thresholds using a three-point difference test, with samples materials for basic taste stimuli used, i.e. reference substances tartaric/citric acid (acidic), quinine hydrochloride/caffeine (bitter), anhydrous sodium chloride (salty), sucrose (sweet), and quercetin/alum (astringent) were used to prepare different tastes and concentrations of liquids. The subjects will then evaluate the appearance (color, texture), taste, flavor, and texture of the six different flavored enteral nutrition preparations. The subjects will then perform manual sensory evaluation of the appearance (color, texture), odor, taste, texture, and other properties of the 6 different flavored enteral nutrition preparations.

DETAILED DESCRIPTION:
1. Combining manual sensory evaluation and electronic bionic sensory, assessing the differences in taste perception between tumor and stroke patients and healthy individuals by measuring the basic taste perception threshold and palatability interval and analyzing facial expressions.
2. Combining manual sensory evaluation with electronic bionic senses and simultaneous facial expression analysis to assess the taste perception characteristics and needs of tumor and stroke patients for different flavors of enteral nutrition preparations.
3. Establishing an information base of electronic tongue taste data, facial expression emotion and flavor data of nutritional preparations based on the electronic tongue and facial expression data of relevant assays obtained simultaneously during the above experiments.

ELIGIBILITY:
Inclusion Criteria:

1. healthy people aged 18-80 years old (including 18 and 80 years old), patients with specific diseases.
2. specific diseases meet the clinical diagnosis criteria and are not in the clinical treatment period (such as radiotherapy or perioperative period)
3. not wearing a denture and having good oral hygiene.
4. normal vision or corrected vision, no hearing impairment, and no mental behavior disorder.
5. voluntarily participate in this trial and sign the informed consent form.

Exclusion Criteria:

1. subjects who may be allergic to the ingredients of the tested food
2. persons who have an aversion to the food to be tasted or who do not consume the food for cultural, ethnic, or other reasons
3. pregnant or lactating women.
4. excessive smokers (>15 cigarettes/day) or heavy drinkers (>25g/day for men and >15g/day for women)
5. Eating disorders (binge eating, anorexia, bulimia nervosa, etc.) and those who cannot eat through the mouth
6. those who underwent ear, nose, and throat, transnasal intracranial occupancy, and oral surgery
7. Those who currently have severe abnormalities of the respiratory system, endocrine system, immune system, nervous system, circulatory system, digestive system, hematopoietic system, and nervous system, and those who have undergone bariatric surgery.
8. currently taking medications that affect the sense of taste
9. Subjects who are participating in other clinical trials.
10. other people who have been determined by the investigator to be unsuitable for participation in this trial, patients with conditions that reduce the likelihood of enrollment or complicate enrollment, such as the presence of conditions that predispose to missed visits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects are healthy people, patients with specific diseases (after radiotherapy for tumors, stroke)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Taste perception threshold | After initial screening and exclusion, subjects who met the inclusion criteria were ready to begin taste threshold testing.
  materials using basic taste stimuli, i.e. reference substances tartaric/citric acid (acid), quinine hydrochloride/caffeine (bitter), anhydrous sodium chloride (salty), sucrose (sweet), quercetin/alum (astringent) to prepare Different flavors and concentrations of solutions were prepared. By the "three-point test", pure water was used as a control to determine the concentration of the flavors caused by The "discrimination threshold" of the sensation was determined by the "three-point test" using pure water as a control.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Chen, Doctor, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Dongcheng district，Peking union medical college hospital, Beijing, Beijing Municipality, China